CLINICAL TRIAL: NCT04231604
Title: Evaluation of a School-based Programme Aimed at Promoting Well-being in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Dublin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: moconnor1
Record Dates: First submitted 2020-01-07; First posted 2020-01-18 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Adolescent Well-Being; Resilience, Psychological

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A Lust for Life programme group (Experimental): A Lust for Life programme will be delivered to adolescents by their school teachers in six weekly lessons. Well-being and resilience will be promoted in each lesson through classroom discussions, videos, classroom activities and homework assignments.
  Interventions: Behavioral: A Lust for Life
- Waiting list control group (Other): Participants will be placed on a twelve-week waiting list for the programme.
  Interventions: Behavioral: Waiting list control

INTERVENTIONS:
Behavioral: A Lust for Life — A Lust for Life is a universal school-based multi-component programme whose target is to build well-being and emotional resilience in adolescents. The programme was informed by evidence-based psychological approaches including mindfulness, cognitive behaviour therapy and positive psychology. It is delivered in six weekly lessons by the adolescents' school teacher and involves classroom discussions, videos, classroom activities and homework assignments.
  Arms: A Lust for Life programme group
Behavioral: Waiting list control — Control group placed on a twelve-week waiting list.
  Arms: Waiting list control group

SUMMARY:
The aim of this pilot study is to evaluate a universal school-based multi-component intervention whose target is to build well-being and emotional resilience in adolescents.

DETAILED DESCRIPTION:
Adolescence is an important developmental phase for prevention and intervention initiatives for well-being and mental health. Accordingly, school has been recommended as an optimal location for such initiatives. Universal programmes - programmes that are designated for all individuals in a population - have a number of advantages, including reducing the risk of stigma and yielding high recruitment rates.

A Lust for Life is a universal school-based multi-component intervention whose target is to build well-being and emotional resilience in adolescents. The programme was informed by evidence-based psychological approaches including cognitive behaviour therapy, positive psychology and mindfulness and consists of six lessons, each delivered by the adolescents' school teacher on a weekly basis. The lessons involve classroom discussions, videos, classroom activities and homework assignments.

Study participants will complete the Adolescent Mental Health Continuum-Short Form, Connor-Davidson Resilience Scale-10, Emotional Literacy and Intervention Inventory-Pupil Checklist, and Mindful Attention Awareness Scale for Children at pre-intervention. Following this, schools randomly assigned to the experimental group will receive A Lust for Life, while those randomly assigned to the control group will be placed on a twelve-week waiting list. The questionnaire measures and a Brief Satisfaction Scale will be completed by participants at post-intervention. In addition, a six-week follow-up assessment will determine whether the effects of the programme are sustained over a period of time. The programme will be delivered in the waiting list control group schools after the six-week follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent
* Enrolled in primary school in Ireland
* Obtain written informed consent from parents/guardians
* Provide written assent

Exclusion Criteria:

* Failure to the meet inclusion criteria

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 604 (Actual)
Dates: Start 2020-01-17 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Well-being measured by the Adolescent Mental Health Continuum-Short Form | 6 weeks after beginning intervention: 19/10/2020
  Scores on the Adolescent Mental Health Continuum-Short Form range from 14 to 84. Higher scores indicate lower well-being.
Well-being measured by the Adolescent Mental Health Continuum-Short Form | 12 weeks after beginning intervention: 01/12/2020
  Scores on the Adolescent Mental Health Continuum-Short Form range from 14 to 84. Higher scores indicate lower well-being.

SECONDARY OUTCOMES:
Resilience measured by the Connor-Davidson Resilience Scale-10 | 6 weeks after beginning intervention: 19/10/2020
  Scores on the Connor-Davidson Resilience Scale-10 range from 0 to 40. Higher scores indicate greater resilience.
Resilience measured by the Connor-Davidson Resilience Scale-10 | 12 weeks after beginning intervention: 01/12/2020
  Scores on the Connor-Davidson Resilience Scale-10 range from 0 to 40. Higher scores indicate greater resilience.

OTHER OUTCOMES:
Emotional literacy measured by the Emotional Literacy and Intervention Inventory-Pupil Checklist | 6 weeks after beginning intervention: 19/10/2020
  Scores on the Emotional Literacy and Intervention Inventory-Pupil Checklist are rated on a four-point scale ranging from 'very like me' to 'not like me at all.' Higher scores indicate higher levels of emotional literacy.
Emotional literacy measured by the Emotional Literacy and Intervention Inventory-Pupil Checklist | 12 weeks after beginning intervention: 01/12/2020
  Scores on the Emotional Literacy and Intervention Inventory-Pupil Checklist are rated on a four-point scale ranging from 'very like me' to 'not like me at all.' Higher scores indicate higher levels of emotional literacy.
Mindfulness measured by the Mindful Attention Awareness Scale for Children | 6 weeks after beginning intervention: 19/10/2020
  Scores on the Mindful Attention Awareness Scale for Children range from 15 to 90. Items are reverse scored so that higher scores indicate higher levels of mindfulness.
Mindfulness measured by the Mindful Attention Awareness Scale for Children | 12 weeks after beginning intervention: 01/12/2020
  Scores on the Mindful Attention Awareness Scale for Children range from 15 to 90. Items are reverse scored so that higher scores indicate higher levels of mindfulness.
Satisfaction with the programme measured by the Brief Satisfaction Scale | 6 weeks after beginning intervention: 19/10/2020
  Scores on each item of the Brief Satisfaction Scale range from 1 to 7. Higher scores indicate greater satisfaction with the programme.

CONTACTS AND LOCATIONS:
Locations (1):
- University College Dublin, Dublin, Leinster, Ireland

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data collected in this research will be archived. Other researchers may contact the investigators to access the de-identified data for use in research into well-being, resilience, emotional literacy and mindfulness.
Time Frame: The data collected in this study will be made available for other researchers after a manuscript reporting on the study's findings has been accepted for publication.
Access Criteria: Data may be accessed for use in research into well-being, resilience, emotional literacy and mindfulness.